CLINICAL TRIAL: NCT03606109
Title: Reducing Hemarthrosis in Tibial Tubercle Osteotomy by the Administration of Intravenous Tranexamic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-00535
Record Dates: First submitted 2018-05-22; First posted 2018-07-30 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Tibial Tubercle Osteotomy
Keywords: Tibial Tubercle Osteotomy; Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Tibial Osteotomy (HTO) (Active Comparator)
  Interventions: Drug: Tranexamic Acid (TXA)
- Tibial Tubercle Ostetomy (TTO) (Active Comparator)
  Interventions: Drug: Tranexamic Acid (TXA)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — One gram of intravenous tranexamic acid (TXA) will be administrated before tourniquet inflation and before closure of the incision, as 1 g has been shown to be a safe amount with minimal side effects

SUMMARY:
The purpose of the proposed study is to evaluate the effects of administering intravenous tranexamic acid (TXA) to patients undergoing high tibial osteotomy (HTO) and tibial tubercle osteotomy (TTO) to minimize hemarthrosis within the knee joint and post operative pain and swelling.

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TTO
* Age 18-60
* Willing and able to provide consent

Exclusion Criteria:

* Legally incompetent or mentally impaired (e.g., minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age
* Older than 60 years of age
* Any patient considered a vulnerable subject
* Have bleeding or clotting disorder
* Preoperative anticoagulation therapy
* Abnormal coagulation profile
* Renal disorder or insufficiency
* Sickle cell disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Alaia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Tibial Osteotomy (HTO) | Tibial Tubercle Ostetomy (TTO)
Started | 31 | 27
Completed | 29 | 26
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Tibial Osteotomy (HTO) | Tibial Tubercle Ostetomy (TTO) | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.65 (8.84) | 34.37 (8.06) | 34.31 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 14 | 13 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29 | 26 | 55

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Blood Loss
Time Frame: Perioperative, up to 2 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Tibial Osteotomy (HTO) | Tibial Tubercle Ostetomy (TTO)
Number analyzed (Participants) | 29 | 26
mL | 67.8 (56.50) | 56.15 (33.92)

2. Secondary Outcome: Score on Visual Analogue Scale (VAS) for Pain
Description: VAS will be used to report post-operative pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Tibial Osteotomy (HTO) | Tibial Tubercle Ostetomy (TTO)
Number analyzed (Participants) | 29 | 26
score on a scale | 7.13 (2.58) | 6.65 (2.66)

3. Secondary Outcome: Score on Visual Analogue Scale (VAS) for Pain
Description: as for outcome 2
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Tibial Osteotomy (HTO) | Tibial Tubercle Ostetomy (TTO)
Number analyzed (Participants) | 29 | 26
score on a scale | 5.82 (1.95) | 5.73 (2.26)

4. Secondary Outcome: Score on Visual Analogue Scale (VAS) for Pain
Description: as for outcome 2
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Tibial Osteotomy (HTO) | Tibial Tubercle Ostetomy (TTO)
Number analyzed (Participants) | 29 | 26
score on a scale | 4.78 (1.76) | 4.77 (2.37)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | High Tibial Osteotomy (HTO) | Tibial Tubercle Ostetomy (TTO)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/27
Other Adverse Events (participants affected / at risk) | 0/31 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03606109/Prot_SAP_000.pdf